CLINICAL TRIAL: NCT07140718
Title: Piloting and Evaluating the Fundamental Adaptive Skills Training (FAST): a New Digitally Augmented Single-Session Transdiagnostic Resilience Intervention
Brief Title: The Fundamental Adaptive Skills Training
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006276
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Fundamental Adaptive Skills Training; Relaxation and Mindfulness Training
Keywords: Transdiagnostic; Digital Mental Health; Resilience

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fundamental Adaptive Skills Training (Experimental)
  Interventions: Behavioral: Fundamental Adaptive Skills Training
- Relaxation and Mindfulness Training (Active Comparator)
  Interventions: Behavioral: Relaxation and Mindfulness Training

INTERVENTIONS:
Behavioral: Fundamental Adaptive Skills Training — The FAST intervention will be approximately 60 minutes in duration. The video component of FAST, animated using the Vyond software, will be presented via computer or projector. Pause points and brief interactive exercises will be added throughout the presentation to promote engagement and ensure comprehension of FAST material. The treatment will be sectioned into thirds: a physical health section focused on sleep hygiene and physical activity, an anxiety sensitivity section dispelling common AS myths, and a social health section. Each section will contain brief psychoeducation focused on dispelling common myths or promoting adaptive skills use.
  Other Names: FAST
  Arms: Fundamental Adaptive Skills Training
Behavioral: Relaxation and Mindfulness Training — The RMT intervention will be primarily psychoeducational and focused on explaining relaxation methods used in various psychological treatments such as progressive muscle relaxation, guided imagery, and mindfulness-focused breathing exercises. Interactive relaxation and mindfulness exercises and brief discussions following each relaxation component will be included to control for time spent on interactive exercises in the FAST condition. The intervention will take approximately 60 minutes. Tailored to control for the effects of general education, practice exercises, and time spent on the FAST intervention, RMT will be a stronger control in comparison to a waitlist or repeated contact condition. Like the FAST intervention, this program will also be digitalized to allow for ease-of-administration.
  Other Names: RMT
  Arms: Relaxation and Mindfulness Training

SUMMARY:
The present study seeks to develop, refine, and test a novel psychological treatment for boosting mental health resilience among college students. This Fundamental Adaptive Skills Training (FAST) will be evaluated in a randomized controlled trial. We will seek to recruit 5 undergraduate students as participants for a pilot phase and 100 undergraduate students for a randomized controlled trial. The primary questions we are seeking to answer in this trial are:

Do participants rate the FAST intervention as acceptable? Does FAST improve sleep quality, physical activity, anxiety sensitivity, loneliness, and social isolation for college students?

Participants will:

Receive the active FAST or a placebo control Relaxation and Mindfulness Training (RMT) and will complete measures at baseline, week 2, and week 4.

DETAILED DESCRIPTION:
The mental health crisis among college students has intensified in recent years, with rising rates of anxiety, depression, and stress. Despite increased institutional efforts, existing mental health services often remain inaccessible or insufficient. The present study proposes and evaluates the Fundamental Adaptive Skills Training (FAST), a novel, single-session intervention designed to promote mental health resilience in college students. FAST will be developed to target empirically supported mechanisms-sleep and physical activity, anxiety sensitivity, loneliness, and social isolation-each linked to a broad range of emotional disorders. Delivered in a digital, group-based format by trained undergraduate peer facilitators, FAST will be scalable, cost-effective, and engaging. This randomized controlled trial will assess the intervention's acceptability and efficacy in improving targeted mechanisms and reducing symptoms of anxiety, depression, and stress over a four-week follow-up period. 100 participants identified as at-risk based on elevated negative affectivity will be randomly assigned to FAST or an active control condition involving mindfulness and relaxation training (RMT). Primary outcomes include improvements in sleep quality, physical activity, anxiety sensitivity, loneliness, and social isolation from baseline through week two and week four follow-up. Similarly, clinical outcomes will include improvements in anxiety, depression, and stress levels as indicators of broader emotional resilience. Findings will advance the science of developing and implementing accessible, evidence-based mental health interventions and may contribute to a novel, scalable solution for addressing mental health issues in higher education settings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* At-risk for emotional disorders as indicated by a PANAS-NA Score >= 20
* Ability to use a computer or smartphone
* Currently enrolled at college/university at the time of study enrollment

Exclusion criteria:

* Adults aged 17 and under
* PANAS-NA Score <= 19
* Inability to use a computer or smartphone
* Not currently enrolled at college/university at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability Questionnaire | Post-intervention through week 4 follow up
  Self report measure indexing intervention acceptability. Scores range from 0 to 27 with higher scores indicating more favorable acceptability.
Athens Insomnia Scale | Baseline through week 4 follow up
  8 item self report measure of sleep quality. Scores range from 0 to 24 with higher scores indicating more severe sleep problems.
Brief Physical Activity Assessment Tool | Baseline through week 4 follow up
  2 item self report measure indexing physical activity. Scores range from 0 to 8 with higher scores indicating more frequent engagement in physical activity.
Anxiety Sensitivity Index 3 | Baseline through week 4 follow up
  18 item self report measure indexing anxiety sensitivity. Scores range from 0 to 72 with higher scores indicating more severe anxiety sensitivity.
UCLA Loneliness 10 | Baseline through week 4 follow up
  10 item self-report measure indexing loneliness. Scores range from 10 to 40 with higher scores indicating more severe loneliness symptoms.
PROMIS Anxiety Scale 8a | Baseline through week 4 follow up
  8 item self report measure of anxiety. Scores range from 8 to 40 with higher scores indicating more severe anxiety symptoms.
PROMIS Depression 8b | Baseline through week 4 follow up
  8 item self report measure indexing depression. Scores range from 8 to 40 with higher scores indicating more severe depression symptoms
Perceived Stress Scale | Baseline through week 4 follow up
  14 item self report measure indexing stress. Scores range from 0 to 56 with higher scores reflecting more severe stress symptoms.

SECONDARY OUTCOMES:
Short Form 12 | Baseline through week 4 follow up
  Quality of life self report measure with 12 items. Scores range from 0 to 100 with higher scores indicating better quality of life

OTHER OUTCOMES:
Positive and Negative Affect Schedule - Negative Affect Scale | Screening through week 4 follow up
  Self report measure indexing negative affectivity. Scores range from 10 to 40 with higher scores indicating worse negative affect.
Demographics | Baseline only
  Self-report demographic questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- FSU Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No